CLINICAL TRIAL: NCT03963765
Title: Transepidermal Application of Metilaminolevulinate in Daylight Photodynamic Therapy in the Treatment of Photodamaged Skin
Brief Title: Transepidermal Application of Metilaminolevulinate in Daylight PDT in the Treatment of Photodamaged Skin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal Fluminense (Other)
Responsible Party: Principal Investigator, Maria Claudia Almeida Issa, Clinical Professor, Universidade Federal Fluminense
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Daylight PDT
Record Dates: First submitted 2019-04-23; First posted 2019-05-28 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Skin Diseases
MeSH Terms: conditions — Skin Diseases | interventions — Lasers, Gas

STUDY DESIGN:
Intervention Model Description: Transepidermic Application of Metilaminolevulinate in Daylight Photodynamic Therapy in the Treatment of Photodamaged Skin
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group I (Standard DL-PDT) (Active Comparator): 1. Superficial skin curettage all face with a dermatological curette
  2. All exposed skin was covered with pure chemical sunscreen
  3. After 15 minutes, a uniform layer of methyl-aminolevulinate (MAL) (Metvix®, Galderma- 1g) was applied to the face without occlusion
  In all protocols, the patients remained indoor for 30 min after procedures and then exposed to daylight in an open environment for 2 hours. After this period, the skin was cleaned with 0.9% saline, and the sunscreen reapplied.
  Interventions: Procedure: Group I (Standard DL-PDT)
- Group II (DL-PDT with microneedles) (Experimental): 1. Superficial skin curettage all face with a dermatological curette
  2. All exposed skin was covered with pure chemical sunscreen
  3. After 15 minutes, a uniform layer of methyl-aminolevulinate (MAL) (Metvix®, Galderma- 1g) was applied to the face without occlusion
  4. A motorized pen with a tip of 17 grouped needles with 0,5mm (Dermapen Beauty®- Korea) was applied without bleeding
  In all protocols, the patients remained indoor for 30 min after procedures and then exposed to daylight in an open environment for 2 hours. After this period, the skin was cleaned with 0.9% saline, and the sunscreen reapplied.
  Interventions: Procedure: Group II (DL-PDT with microneedles)
- Group III (DL-PDT with CO2 laser) (Experimental): 1. Superficial skin curettage all face with a dermatological curette
  2. All exposed skin was covered with pure chemical sunscreen
  3. After 15 minutes and removing excess sunscreen, Ablative Fractional Laser (AFXL), CO2 laser, roller-type ferrule, composed of one row with seven fractionating pins (7x1), 60 W, 15 mJ/pixel, 125μm/pixel, 2 mm spacing between ablation zones, density <1% (Pixel Alma Lasers ®) was applied, single-pass
  4. A uniform layer of methyl-aminolevulinate (MAL) (Metvix®, Galderma- 1g) was applied to the face without occlusion
  In all protocols, the patients remained indoor for 30 min after procedures and then exposed to daylight in an open environment for 2 hours. After this period, the skin was cleaned with 0.9% saline, and the sunscreen reapplied.
  Interventions: Procedure: Group III (DL-PDT with CO2 laser)
- Group IV (DL-PDT with microdermabrasion) (Experimental): 1. Superficial skin curettage all face with a dermatological curette
  2. Microdermabrasion with aluminum oxide crystal (Pan Eletronic®) was performed after superficial skin curettage. Three passes on the skin in different directions (vertical, horizontal, and oblique) were applied
  3. All exposed skin was covered with pure chemical sunscreen
  4. After 15 minutes, a uniform layer of methyl-aminolevulinate (MAL) (Metvix®, Galderma- 1g) was applied to the face without occlusion
  In all protocols, the patients remained indoor for 30 min after procedures and then exposed to daylight in an open environment for 2 hours. After this period, the skin was cleaned with 0.9% saline, and the sunscreen reapplied.
  Interventions: Procedure: Group IV (DL-PDT with microdermabrasion)

INTERVENTIONS:
Procedure: Group I (Standard DL-PDT) — Daylight photodynamic therapy with photosensitizer (MAL - Metvix, Galderma ®)
  Other Names: Daylight PDT
  Arms: Group I (Standard DL-PDT)
Procedure: Group II (DL-PDT with microneedles) — Daylight photodynamic therapy with photosensitizer (MAL - Metvix, Galderma ®) and Microneedles - motorized pen with a tip of 17 grouped needles with 0,5mm (Dermapen Beauty®- Korea) as a techniques of transepidermal drug delivery (TED)
  Other Names: Daylight PDT with microneedles
  Arms: Group II (DL-PDT with microneedles)
Procedure: Group III (DL-PDT with CO2 laser) — Daylight photodynamic therapy with photosensitizer (MAL - Metvix, Galderma ®) and Ablative Fractional Laser (AFXL), CO2 laser, roller-type ferrule, composed of one row with seven fractionating pins (7x1), 60 W, 15 mJ/pixel, 125μm/pixel, 2 mm spacing between ablation zones, density <1% (Pixel Alma Lasers ®) was applied, single-pass
  Other Names: Daylight PDT with CO2 laser
  Arms: Group III (DL-PDT with CO2 laser)
Procedure: Group IV (DL-PDT with microdermabrasion) — Daylight photodynamic therapy with photosensitizer (MAL - Metvix, Galderma ®) and Microdermabrasion - aluminum oxide crystal (Pan Eletronic®) as a techniques of transepidermal drug delivery (TED)
  Other Names: Daylight PDT with microdermabrasion
  Arms: Group IV (DL-PDT with microdermabrasion)

SUMMARY:
Chronic sun exposure enhances the incidence of cutaneous neoplasms (NMSC - non melanoma skin cancer), wrinkles, roughness, telangiectasia and irregular pigmentation of the skin. Nowadays, actinic keratosis (AK) are considered in situ squamous cell carcinoma (SCC), and should be managed that way. Conventional topical Photodynamic therapy (PDT) has proven its efficacy on treatment of AK and cancerization field. PDT's action in global improvement of photodamaged skin, texture, pigmentation and reduction of wrinkles has been well documented in literature. Immunohistochemical and histopathological essays describe the hypothesis of conventional PDT's mechanisms of action in photoaging by dermal remodeling, with enhancement of collagen, statiscally significant. Daylight-Photodynamic Therapy (DL-PDT) is a new modality that keeps the efficacy of topical PDT in treatment of AK and cancerization field, but painless and more practically. Until this moment, there is no report of DL-PDT efficacy on photorejuvenation and actinic keratosis evaluated by clinical, histopathological and immunohistochemical studies. The investigator's aim is to evaluate the alterations induced by isolated DLPDT or DLPDT associated with other techniques of transepidermal drug delivery (microneedles, CO2 laser and microdermabrasion) in the treatment of field cancerization in photodamaged skin with actinic keratosis, through clinical evaluation, histopathological and immunohistochemical studies. It is an interventional, prospective, randomized controlled, parallels-groups, four-arm trial with 1:1 allocation ratio study performed in forty patients attended at the Dermatology Service of Hospital Universitário Antonio Pedro- Universidade Federal Fluminense.

DETAILED DESCRIPTION:
This is a randomized controlled, parallels-groups, four-arm trial with 1:1 allocation ratio study on the clinical, histological and immunohistochemical changes induced by Daylight-Photodynamic Therapy (DL-PDT) in 40 patients presenting face-photodamaged skin with actinic keratosis, attended at the Dermatology outpatient clinic of Hospital Antônio Pedro (HUAP) of Universidade Federal Fluminense - UFF, who meet the inclusion criteria and agree to sign the informed consent form (TCLE) for participation in clinical research. There will be four treatment groups with different protocols. These protocols were chosen by hand draw using two boxes containing folded papers. One with the 4 numbers of the groups (1, 2, 3, 4), and another with 4 papers with the names of the protocols. At each draw, one paper from each box was withdrawn, and the combined results from the two boxes defined the treatments of each group. Group I was randomly selected to be DL-PDT alone (standard procedure - group control); Group II was randomly selected to be DL-PDT with TED (microneedles); Group III was randomly selected to be DL-PDT with TED (CO2 laser) and Group IV was was randomly selected to be DL-PDT with TED (microdermabrasion with crystal peeling). Two treatment sessions will be performed with a 4-week interval, regardless of the protocol chosen per group. Patients will be numbered according to the registration for participation in the study. These numbers will be distributed in 4 groups randomly through the computer, using an Apple application called Random (random number generator: seller Mireia Lluch Ortoloa, category utilities, version 1). Each DL-PDT session will consist of: superficial skin curettage all face with a dermatological curette; application of pure chemical sunscreen for 15 minutes; application of methyl-aminolevulinate (Metvix®, GALDERMA), approved by ANVISA under Registration No. 1291600650016, for 30 minutes without occlusion, before exposure to daylight for 2 hours. Regarding the association of techniques, these will be varied according to the group. For clinical evaluation, patient data will be recorded on the evaluation form, and photographs with the same position and lighting patterns will be performed before and after predetermined periods. For histological and immunohistochemical evaluations, skin biopsies will be performed before and after 3 months of the last treatment session.

ELIGIBILITY:
Inclusion Criteria:

* Both gender;
* Fitzpatrick phototypes I - IV;
* age between 40 and 75 years;
* photodamaged skin with at least 1 lesion of actinic keratosis

Exclusion Criteria:

* Pregnancy and lactation;
* photosensitivity;
* smoking;
* malignant neoplasms;
* infections;
* immunosuppression;
* collagenoses;
* any systemic disease or emotional/psychological disorder that could contraindicate the procedure.
* any topical treatment or interventions for at least three months before the study started

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-02-03 (Actual); Primary Completion 2018-12-05 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Quantitative clinical evaluation of Actinic keratoses | 6 months
  Numbers of Actinic keratoses on the face: count of lesions before treatment and one month/three months/six months after the second session.
Qualitative clinical evaluation of Actinic keratoses | 6 months
  Actinic keratoses will be classified by degrees of thickness (grades 1, 2 and 3), based on the Olsen scale (J Am Acad Dermatol. 1991 May;24(5 Pt 1):738-43), before treatment and one month/three months/six months after the second session.
Qualitative evaluation of global clinical skin change | 6 months
  The overall improvement of photodanificated skin was evaluated using the GAIS scale (Global Aesthetic Improvement Scale) which ranges from: 1 = very much improvement; 2 = marked improvement; 3 = improved; 4 = no change; 5 = worse. Also performed before treatment and one month/three months/six months after the second session.

SECONDARY OUTCOMES:
Histological evaluation: Routine stain - haematoxylin and eosin | 1 year
  Morphologic study: the aspect of the corneal layer and epidermis, the thickness of the epidermis (distance between granular layer and basal layer), the extension of the keratinocytes atypia, the amount and cytological aspect of melanocytes, the thickness of the subepidermal collagen (distance between membrane basal and onset of solar elastosis in the papillary dermis), distribution of solar elastosis (diffuse or compact distribution), the presence and the type of inflammatory infiltrate, the presence or absence of ectasia in the papillary dermis vessels. These measurements were performed through an ocular lens with a millimeter ruler (Olympus).
Histological evaluation: Special stains (Orcein and Picrosirius) | 1 year
  Orcein (morphologic study): the distribution of solar elastosis and the organization of the elastic fibers (elaunin and oxytalan fibers present in the papillary dermis and dermo-epidermal junction).
  Picrosirius (morphometry of dermis collagen)
Immunohistochemistry: epidermis and dermis | 1 year
  Expression of these substrates:
  Ki 67, P53 (wild type and mutated): percentage and extent (1/3, 2/3 or 3/3) in the epidermis
  Collagen type I and III, MMP 1,3,9, TIMP 1: semiquantitative method: 0, absence of expression; +, weak expression; ++, moderate expression; +++, strong expression.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Claudia Issa, Principal Investigator — Professor
Locations (1):
- Hospital Universitário Antonio Pedro - Universidade Federal Fluminense, Niterói, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No